CLINICAL TRIAL: NCT03760380
Title: Pilot Study: Comparing Pain and Kinematic Outcomes of Two Gait-Modifying Shoe Interventions on Knee Osteoarthritis Acutely and Over a 12 Week Period
Brief Title: Comparing Pain and Kinematic Outcomes of Two Gait-Modifying Shoe Interventions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor funding shortage
Sponsor: University of Florida (Other)
Collaborators: Scientific Motion Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: OCR17682
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Arthritis Knee
Keywords: osteoarthritis (OA); gait modifying shoe
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Phase 1 All subjects will perform the same procedures with all the experimental interventions (Sole 1 - Neutral, Sole 1--Offset, Sole 2 - Neutral, Sole 2 - Offset)
  Phase 2 Subjects will be assigned one of two shoes/soles (either Sole 1-Offset or Sole 2- Offset) for home use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Phase 1 Short Term (Experimental): Participants will serve as their own control. Questionnaires and gait measures will be collected during an initial visit using the experimental shoe device. All subjects will perform the same procedures with all the experimental interventions (Sole 1 - Neutral, Sole 1--Offset, Sole 2 - Neutral, Sole 2 - Offset)
  Interventions: Device: Sole 1 - Neutral; Device: Sole 1 - Offset; Device: Sole 2 - Neutral; Device: Sole 2 - Offset
- Phase 2 Long Term (Experimental): Participants will serve as their own control. Questionnaires, balance, functional and gait measures will be collected during four different visits over a twelve week period (once at baseline visit, 4, 8, and 12 week visits) using the experimental shoe device. Patients will also complete a home walking program using the shoe device over the twelve week period. Subjects will be assigned one of two shoes/soles (either Sole 1-Offset or Sole 2- Offset) for home use.
  Interventions: Device: Sole 1 - Offset; Device: Sole 2 - Offset

INTERVENTIONS:
Device: Sole 1 - Neutral — Appropriately-designed, stimulatory - but not mechanically supportive -device to enhance control of balance, postural sway and key features of walking gait in arthritic knee patients. The gait-modifying shoes will initially be neutrally aligned to create the smallest amount of instability. This is defined as the location which creates the smallest amount of instability.
  Arms: Phase 1 Short Term
Device: Sole 1 - Offset — Appropriately-designed, stimulatory - but not mechanically supportive -device to enhance control of balance, postural sway and key features of walking gait in arthritic knee patients. The offset sole will be placed in a position that may reduce the knee adduction moment. The anterior elements will be placed 1 cm medially from the neutral position and the posterior pod will be moved 1 cm laterally from the neutral position.
Device: Sole 2 - Neutral — Appropriately-designed, stimulatory - but not mechanically supportive -device to enhance control of balance, postural sway and key features of walking gait in arthritic knee patients. The gait-modifying shoes will initially be neutrally aligned to create the smallest amount of instability.This is defined as the location which creates the smallest amount of instability.
  Arms: Phase 1 Short Term
Device: Sole 2 - Offset — Appropriately-designed, stimulatory - but not mechanically supportive -device to enhance control of balance, postural sway and key features of walking gait in arthritic knee patients. The offset sole will be placed in a position that may reduce the knee adduction moment. The anterior elements will be placed 1 cm medially from the neutral position and the posterior pod will be moved 1 cm laterally from the neutral position.

SUMMARY:
This study involves the use of a newly designed shoe device for knee arthritis patients that may help reduce knee pain and improve function.

DETAILED DESCRIPTION:
This study involves the use of a newly designed shoe device for knee arthritis patients that may help reduce knee pain and improve function. This is a 2-phase study designed to evaluate knee pain and function in healthy participants with a history of medial knee arthritis.

The purpose of this study is to evaluate: 1. how using the shoe device will affect a person's walking gait and balance over a single day; and 2. how using the shoe device over the course of a 12-week period will affect a person's walking gait and balance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic, OA-related knee pain
* Diagnosis of medial compartment knee OA (unilateral or bilateral)
* Moderate pain of ≥4 out of 10 points while performing a weight-bearing activity
* Kellgren and Lawrence score of 2, 3, or 4 evidenced on routine, standard-of-care x-ray within the last 2 years prior to enrollment
* Able to walk unassisted for at least 10 minutes at a time
* Wear a Women's shoe size of 6.5 to 13 or a Men's shoe size of 5 to 12.

Exclusion Criteria:

* Patients suffering from acute septic or inflammatory arthritis
* Unstable cardiovascular, orthopaedic, or neurological conditions, uncontrolled diabetes, or any condition that would preclude exercise in moderate duration, moderate workload trials
* Received a corticosteroid injection or invasive procedures within prior 6 months of the study
* History of avascular necrosis in the knee
* History of knee buckling
* Joint replacement in any lower extremity joint that has not optimally recovered (e.g. still causes significant pain or affects mobility) as determined by the PI.
* Experienced more than 3 falls within the last year
* Currently using any knee brace on a regular basis for the knee pain, with the exception of basic knee sleeves
* Pathological osteoporotic fracture
* Severe symptomatic degenerative arthritis in lower limb joints other than the knees
* Severe back pain, prior spinal fusion or spinal deformity that would affect gait
* Major cardiac or pulmonary conditions and any orthopedic limitation that precludes their ability to independently walk for 10 minutes or longer
* Knee flexion contracture greater than 15°
* Knee flexion of less than 90°
* Any major injury to either knee within the prior 12 months
* Currently enrolled in a supervised physical therapy program

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-16 (Estimated); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Change in NRS pain (Pain Numeric Rating Scale) score. | Baseline (Phase 1); Baseline (Phase 2), Week 4, Week 8, Week 12
  Participants selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as one can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
Change in WOMAC (Western Ontario and McMaster Universities Arthritis Index) score | Baseline (Phase 2), Week 4, Week 8, Week 12
  Self-administered questionnaire consisting of 24 items divided into 3 subscales [total score 0-96; subscales from 0-20 (pain)/0-8(stiffness)/0-68(physical function)]. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
Change in SF-36 disability score. | Baseline (Phase 2), Week 4, Week 8, Week 12
  Eight scaled scores, where each scale is directly transformed into a 0-100 scale. The lower the score the more disability.
Change in Timed Up & Go (TUG) Test score. | Baseline (Phase 2), Week 4, Week 8, Week 12
  Time it takes for participant to rise from chair, walk 3 meters, turn around, walk back and sit down.
Change in Stair Climb time score. | Baseline (Phase 2), Week 4, Week 8, Week 12
  Time it takes participant to walk up on flight of stairs (12 steps).

CONTACTS AND LOCATIONS:
Overall Officials: Hari K Parvataneni, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No